CLINICAL TRIAL: NCT06146322
Title: Barley Beta-glucan, Glycemic Control, and Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Responsible Party: Principal Investigator, Martine Perrigue, Assistant Professor, Nutrition and Exercise Physiology, Washington State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 17735
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Diet, Healthy; Blood Sugar; High; Diabetes; Appetite and General Nutritional Disorders; Appetitive Behavior
Keywords: Beta-glucan; Fiber; Glycemic Control; Appetite
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus; Appetitive Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: WR — Unsweetened preload condition: 240 mL white glutinous rice, 250 kcal, 0 g β-glucan
Other: LB — Unsweetened preload condition: 240 mL low β-glucan barley, 250 kcal, ~4 g β-glucan
Other: MB — Unsweetened preload condition: 240 mL medium β-glucan barley, 250 kcal, ~5 g β-glucan
Other: HB — Unsweetened preload condition: 240 mL high β-glucan barley, 250 kcal, ~6 g β-glucan
Other: WR+50g HFCS — Sweetened condition with high fructose corn syrup (HFCS): 240 mL white glutinous rice + 50g HFCS, 391 kcal, 0 g β-glucan
Other: LB + 50 g HFCS — Sweetened condition with high fructose corn syrup (HFCS): 240 mL low β-glucan barley + 50 g HFCS, 391 kcal, ~4 g β-glucan
Other: MB + 50 g HFCS — Sweetened condition with high fructose corn syrup (HFCS): 240 mL medium β-glucan barley + 50 g HFCS, 391 kcal, ~5 g β-glucan
Other: HB + 50 g HFCS — Sweetened condition with high fructose corn syrup (HFCS): 240 mL high β-glucan barley + 50 g HFCS, 391 kcal, ~6 g β-glucan

SUMMARY:
Novel barley varieties high in the soluble fiber β-glucan have the capacity to improve population health through improving glycemic control. Sweetened and unsweetened wholegrain barley foods were tested in a randomized, controlled, crossover human clinical trial to assess impact on postprandial appetite and food intake.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age
* Body Mass Index (BMI) values of 18.5-40.0 kg/m2
* Normal fasting blood glucose (<100 mg/dL)

Exclusion Criteria:

* Use of medications known to be associated with weight change (e.g., beta-blockers)
* Use of steroid pills or shots such as prednisone or cortisone
* Use of nicotine
* Weight change of ten or more pounds in the last three months
* Major daily variation in physical activity (e.g., athletes in training)
* History of extensive small bowel surgery or surgery to treat obesity
* History of heart attack, stroke, or bypass
* History of cancer within the last five years (exception: non-melanoma skin cancer)
* Recent or current medical diagnosis or medical treatment that would alter appetite, energy needs, satiety, and/or could impact the results of the trial
* Medical diagnoses of diabetes, cardiovascular disease, high levels of blood lipids, asthma, cold, and flu (exception: hypertension, if treated with medication prescribed more than three months prior to the screening activity)
* Fear of blood or needles
* Dietary restrictions that would interfere with consuming test foods (e.g., gluten intolerance, vegan, corn syrup allergy)
* Following a weight modification diet
* Sensitive to food textures present in the test foods
* Following personal schedules that would not permit attendance at all scheduled testing sessions
* Unable to comprehend the nature of the trial or instructions
* Unable to understand English sufficiently to complete the trial

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Postprandial glycemic response | 4 hours
  Blood glucose measured every 15 minutes post-preload ingestion
Subjective appetite | 4 hours
  Self-reported appetite measured using Visual Analogue Scale (VAS) every 15 minutes post-preload ingestion
Food intake | 30 minutes
  Food intake at a 16-item ad libitum test meal served 4 hours post-preload ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Martine Perrigue, PhD, RDN, Principal Investigator — Washington State University
Locations (1):
- Washington State University, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No